CLINICAL TRIAL: NCT02690090
Title: Phase 4 Study Determining the Safety of Enoxaparin Prophylaxis in Critically Ill Adults With Severe Renal Insufficiency
Brief Title: Safety Study of Enoxaparin Prophylaxis in Critically Ill Adults With Severe Renal Insufficiency
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Enox-TOH-0001-RP
Record Dates: First submitted 2014-01-10; First posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Hemorrhage
Keywords: Deep Vein Thrombosis; Prophylaxis; Critically ill adults
MeSH Terms: conditions — Hemorrhage; Venous Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- enoxaparin: enoxaparin prophylaxis as directed by treating Intensivist

SUMMARY:
The investigators study is the first step (a pilot study) in determining whether the manufacturer's recommended dose of a blood thinner called enoxaparin, in adults who are patients in an intensive care unit and have severely reduced kidney function (less than or equal to approximately 30% of their normal function) is safe with respect to the adverse effect of bleeding.

The investigators hypothesis is that studying these patients, going forward in time, without interfering with their care, to eventually determine if this blood thinner is safe at reduced doses, is feasible.

DETAILED DESCRIPTION:
Objectives:

To determine the feasibility of conducting a single centre, open-label, prospective study to inform preparation for a prospective phase III study evaluating the efficacy & safety of enoxaparin prophylaxis in critically ill adults with creatinine clearance < 30 mL/min.

Study Design:

A pilot open-label, single-arm, prospective study.

Patients:

Critically ill adults (> 18 years) with creatinine clearance < 30 mL/min.

Setting:

The Ottawa Hospital Intensive Care Units

Sample Size: n=30.

Intervention:

Study patients will receive enoxaparin 30 mg S.C. daily for VTE prophylaxis as directed by their responsible Intensivist. The investigators are not directing this clinical intervention in any manner.

Primary/Feasibility Outcomes: screening and enrolment rates with a goal of recruiting at least 5 patients collectively, from both ICUs, per month.

Secondary/Clinical Outcomes: Determining the accumulation of anti-Xa concentrations, if any, recording of the rates of major bleeding, VTE, and HIT during the study.

Trial Duration:

Anticipated 24 months.

Analysis:

Statistical analysis will be performed using SAS software through the Ottawa Hospital Methods Centre. Patient demographics and clinical baseline characteristics will be described. Continuous variables will be presented as mean (SD), ordinal variables as medians (IQR) and categorical variables as proportions. Cox proportional hazards analysis will be used to evaluate an association between trough anti-Xa levels and major bleeding.

ELIGIBILITY:
Inclusion Criteria:

* body weight ≥ 45 kg
* expected ICU length of stay ≥ 72 hours
* severe renal insufficiency, defined by calculated creatinine clearance (CrCl) < 30 mL/min using the Cockcroft-Gault formula
* All patients with severe renal insufficiency at ICU admission will be included, regardless of chronicity of renal disease. This includes patients with pre-existing dialysis dependence via intermittent hemodialysis and peritoneal dialysis; patients with acute kidney injury requiring SLED (sustained low-efficiency dialysis) will also be included.

Exclusion Criteria:

* neurological surgery in last 3 months
* epidural catheter insertion within previous 12 hours
* ICU admission > 2 weeks
* receipt of > 2 doses of LMWH while in ICU or in hospital within 7 days prior to study enrolment
* active bleeding; platelet count < 50 x 109/L
* INR or aPTT > 2 times the upper limit of normal
* need for therapeutic anticoagulation; previous adverse reaction to heparin based products
* contraindication to blood product transfusion
* pregnant or lactating women
* life expectancy < 2 weeks or receiving palliative care
* previous enrolment in current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult critically ill patients with creatinine clearance < 30 mL/min and requiring thromboprophylaxis during their ICU course.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-03 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Determine the rate of patient enrollment into this study within the 24 month allotted time frame of recruitment | 24 months
  This is a pilot feasibility study

SECONDARY OUTCOMES:
Measure bioaccumulation of Enoxaparin, if any, defined as at least one trough anti-Xa level measuring > 0.4 IU/mL | 24 hours
  Trough Anti-Xa concentration at baseline, 4, 8, 12, 16 & 24 hours of ICU day 1
Record incidence of major bleeding episodes using the HEME bleeding assessment tool | Daily until ICU discharge or a maximum of the first 10 days of ICU stay, whichever is less
Record incidence of VTE | Daily until ICU discharge or a maximum of the first 10 days of ICU stay, whichever is less
Measure bioaccumulation of Enoxaparin, if any, defined as at least one trough anti-Xa level measuring > 0.4 IU/mL | ICU stay until discharge or a maximum of the first 10 days of ICU stay, whichever is less
  Trough Anti-Xa concentration will be measured on days; 2, 3, 4, 7 & day of ICU discharge or ICU day 10, whichever is less

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh V Patel, MD PharmD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No